CLINICAL TRIAL: NCT03078413
Title: Late Function After Surgery for Transposition of the Great Arteries
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Eric Ebenroth, Clinical Associate Professor of Pediatrics, Indiana University
Other Study IDs: 1011003175
Record Dates: First submitted 2017-03-02; First posted 2017-03-13 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Transposition of Great Vessels
Keywords: Mustard Procedure
MeSH Terms: conditions — Transposition of Great Vessels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators proposed to review the exercise tolerance, cardiac function, and quality of life in patients born with transposition of the great arteries that have undergone surgery with either the Mustard or Senning procedure. Participants will complete a questionnaire. The investigators will review the participants' recent cardiac function testing which will assess their current health status. These tests include an echocardiogram, a metabolic exercise stress test, cardiac imaging, and a 24-hour Holter monitor. This collection of testing results will be compared specifically with previously acquired data during the first phases of this study (published in 2001 and 2007).

DETAILED DESCRIPTION:
1. Enrolled subjects must consent to the study and authorize release of health information. All studies obtained as part of this research study are considered part of routine care.
2. Prior to testing, subjects must complete a questionnaire assessing quality of life. This is the same questionnaire that has been used in the previous portions of this study.
3. The investigators will review results of cardiac imaging for all participants consisting of a cardiac MRI or cardiac CT obtained within the last 5 years. If this data does not exist or is outdated, participants will have a new study.
4. The investigators will review results of cardiac imaging for all participants consisting of an echocardiogram within the last 5 years. If this data does not exist or is outdated, participants will have a new study.
5. The investigators will review results of cardiac function testing for all participants consisting of an exercise stress test obtained within the last 5 years. If this data does not exist or is outdated, participants will have a new study. End criteria for the exercise stress test includes either

   a. Achieving two or more of the following: i. Heart rate of > 95% of age-predicted maximum (using equation 220-age = maximal heart rate) ii. RER > 1.1 iii. VO2 plateau defined as The VO2 plateau was defined as a change in VO2 during the final minute of exercise less than 2 SD below the mean of increases between previous workloads iv. RPE > 8 on OMNI RPE scale v. Volitional exertion OR b. Achievement of any of the contraindications to exercise testing.
6. The investigators will review results of cardiac rhythm monitoring for all participants consisting of a 24 hour Holter monitor obtained within the last 5 years. If this data does not exist or is outdated, participants will have a new study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have had an atrial switch procedure (Mustard or Senning operation). Since these operations were last performed on this population in the early 1980's all patients will be older than 18 years of age at the time of enrollment.
2. Patients must be willing to adhere to the guidelines of this study

Exclusion Criteria:

1. Patients who are medically unstable
2. Patients that are non-ambulatory
3. Patients with a history of exercise induced arrhythmia
4. Patients with atrial flutter or history of treatment resistant atrial flutter
5. Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must have had an atrial switch procedure (Mustard or Senning operation) and have participated in the prior two installments of this study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Survival | 2 years
  Survival following Mustard procedure to time of study

SECONDARY OUTCOMES:
Quality of Life | 2 years
  QOL as assessed by questionnaire
Exercise Capacity | 2 years
  Peak oxygen consumption in mL/kg/min
Cardiac Function | 2 years
  RV ejection fraction (%) as measured by echocardiogram and MRI/CT
Cardiac rhythm assessment | 2 years
  Percentage of abnormal rhythm

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martins P, Castela E. Transposition of the great arteries. Orphanet J Rare Dis. 2008 Oct 13;3:27. doi: 10.1186/1750-1172-3-27. PMID 18851735
- [Background] Moons P, Gewillig M, Sluysmans T, Verhaaren H, Viart P, Massin M, Suys B, Budts W, Pasquet A, De Wolf D, Vliers A. Long term outcome up to 30 years after the Mustard or Senning operation: a nationwide multicentre study in Belgium. Heart. 2004 Mar;90(3):307-13. doi: 10.1136/hrt.2002.007138. PMID 14966055
- [Background] Warnes CA. Transposition of the great arteries. Circulation. 2006 Dec 12;114(24):2699-709. doi: 10.1161/CIRCULATIONAHA.105.592352. PMID 17159076
- [Background] Dos L, Teruel L, Ferreira IJ, Rodriguez-Larrea J, Miro L, Girona J, Albert DC, Goncalves A, Murtra M, Casaldaliga J. Late outcome of Senning and Mustard procedures for correction of transposition of the great arteries. Heart. 2005 May;91(5):652-6. doi: 10.1136/hrt.2003.029769. PMID 15831655
- [Background] Ebenroth ES, Hurwitz RA. Functional outcome of patients operated for d-transposition of the great arteries with the Mustard procedure. Am J Cardiol. 2002 Feb 1;89(3):353-6. doi: 10.1016/s0002-9149(01)02242-1. No abstract available. PMID 11809443